CLINICAL TRIAL: NCT01694004
Title: Duodenal Lipid Sensing and Nutrient Absorption
Brief Title: Nutrient Sensing in the Duodenum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Robyn Tamboli, Research Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #121111; P30DK058404 (NIH)
Record Dates: First submitted 2012-09-24; First posted 2012-09-26 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: The Effect of LCFA on Nutrient Absorption
Keywords: Nutrient absorption; Duodenal feeding tube; Gut-brain-gut axis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Benzocaine Infusion into Duodenum (Experimental): The investigator will conduct a study in 20 lean (BMI = 19-27 kg/m2) subjects involving intravenous (IV) and intraduodenal (ID) infusions of glucose tracers or amino acid traces and measurement of tracer rate of appearance in the plasma. An ID infusion of LCFA will allow the investigators to determine if LCFA can alter nutrient absorption and glucose and amino acid metabolism. Benzocaine will be added to the ID infusion of LCFA to inhibit nerve terminals in the duodenum thereby preventing gut-brain communication. Plasma levels of glucose and amino acid tracers, glucose oxidation (13CO2 breath test), gut hormones (CCK, GIP, PYY, GLP-1, ghrelin), and bioactive lipids (N-acyl phosphatidylethanolamines, NAPEs) will be measured during all infusion periods.
  Interventions: Drug: Benzocaine Infusion into Duodenum

INTERVENTIONS:
Drug: Benzocaine Infusion into Duodenum

SUMMARY:
Preliminary studies in humans suggest that the presence of lipids in the gut can modify glucose absorption. The overall hypothesis of this proposal is that long chain fatty acid sensing in the duodenum has a significant role in modifying nutrient (glucose and amino acid) absorption from the GI tract through a gut-brain-gut axis.

DETAILED DESCRIPTION:
The investigator will conduct a study in 20 lean (BMI = 19-27 kg/m2) subjects involving intravenous (IV) and intraduodenal (ID) infusions of glucose tracers or amino acid tracers and measurement of tracer rate of appearance in the plasma. An ID infusion of LCFA will allow the investigators to determine if LCFA can alter nutrient absorption and glucose and amino acid metabolism. Benzocaine will be added to the ID infusion of LCFA to inhibit nerve terminals in the duodenum thereby preventing gut-brain communication. Plasma levels of glucose and amino acid tracers, glucose oxidation (13CO2 breath test), gut hormones (CCK, GIP, PYY, GLP-1, ghrelin), and bioactive lipids (N-acyl phosphatidylethanolamines, NAPEs) will be measured during all infusion periods.

ELIGIBILITY:
Inclusion Criteria:

* BMI = 19-27 kg/m2
* 30-55 years of age

Exclusion Criteria:

* Contraindication for nasal tube placement (e.g. deviated septum, prior upper gastrointestinal bleed, or history of easy bleeding)
* Prior gastric or intestinal surgery or pancreas resection
* Females with a positive pregnancy test
* Known history of intestinal diseases including (but not limited to) inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), celiac sprue, Barrett's esophagus
* Type 1 or type 2 diabetes
* Gastroenteritis (diarrhea and/or vomiting) or constipation within the past week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-10-27 (Actual); Study Completion 2014-10-27 (Actual)

PRIMARY OUTCOMES:
Nutrient Absorption | 6 hours
  Stable isotope tracers (glucose or amino acid) will be administered intravenously (IV) and intraduodenally (ID) and tracer rate of appearance in the plasma will be measured.

SECONDARY OUTCOMES:
Substrate Oxidation | 6 hours
  Oxidation of intraduodenally administered glucose or amino acid will be determined by the amount of 13C recovered from expired air.
Gut Hormone Levels | 6 hours
  Plasma levels of gut hormones will be measured by standard RIA or ELISA assays

OTHER OUTCOMES:
Bioactive Lipids | 6 hours
  Plasma levels of N-acyl phosphatidylethanolamines (NAPES)will be measured by LC-MS

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Tamboli, PhD, Principal Investigator — Vanderbilt University Medical Center; Naji Abumrad, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided